CLINICAL TRIAL: NCT03229486
Title: A Prospective, Double-blind, Randomized Study to Investigate the Effect of Sugammadex vs. Neostigmine/Glycopyrrolate on Emergence Delirium During Sevoflurane-rocuronium Anesthesia in Pediatric Patients
Brief Title: Effect of Sugammadex vs. Neostigmine/Glycopyrrolate on Pediatric Emergence Delirium in Sevoflurane-rocuronium Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Tae-Kyun Kim, Associate professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PusanNUYH
Record Dates: First submitted 2017-06-29; First posted 2017-07-25 (Actual); Results first posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Emergence Delirium
Keywords: emergence delirium; tonsillectomy
MeSH Terms: conditions — Emergence Delirium | interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sugammadex Injection [Bridion] (Experimental): reversal of neuromuscular blockade with sugammadex
  Interventions: Drug: Sugammadex Injection [Bridion]
- Neostigmine+Glycopyrronium (Active Comparator): reversal of neuromuscular blockade with neostigmine & glycopyrrolate
  Interventions: Drug: Neostigmine+Glycopyrronium

INTERVENTIONS:
Drug: Sugammadex Injection [Bridion] — Return to T2 point (two contractions) on TOF device is replied by iv 2 mg/kg sugammadex administration, contained in a blinded syringe.
  Other Names: Sugammadex
  Arms: Sugammadex Injection [Bridion]
Drug: Neostigmine+Glycopyrronium — Return to T2 point (two contractions) on TOF device is replied by iv 0.06 mg/kg neostigmine and 0.005 mg/kg glycopyrrolate administration, contained in a blinded syringe.
  Other Names: Neostigmine
  Arms: Neostigmine+Glycopyrronium

SUMMARY:
The aim of this study is to investigate the effect of sugammadex vs. a conventional acetylcholinesterase inhibitor, neostigmine on emergence delirium (ED) during sevoflurane-rocuronium anesthesia in pediatric patients Additionally, the efficacy features of sugammadex compared to neostigmine will be examined by measuring the time from start of administration of reversal agents to recovery of train-of-four (TOF) ratio to 0.7, 0.8, and 0.9.

Although the etiology of ED remains unclear, a sense of suffocation or breathing difficulty during emergence from anesthesia has been suggested as a possible cause. Thus, reversal of neuromuscular blockade with sugammadex in pediatric patients maintained with sevoflurane-rocuronium anesthesia may decrease ED due to its faster reversal of neuromuscular blockade and decreased possibility of residual blockade.

DETAILED DESCRIPTION:
Emergence delirium (ED) is a postanesthetic phenomenon that develops in the early phase of general anesthesia recovery, (usually within the first 30 minutes,) and is defined as "a disturbance in a child's awareness of and attention to his/her environment with disorientation and perceptual alterations including hypersensitivity to stimuli and hyperactive motor behavior" . Children are often irritable, uncompromising, uncooperative, incoherent, and inconsolably crying, moaning, kicking, or thrashing. The incidence of ED varies from 2 to 80%, occurring more frequently in preschool boys. Risk factors also include the following: sevoflurane or desflurane anesthesia; ear, nose and throat surgery; preoperative anxiety. ED is known to increase physical, psychological, and financial burdens in the postanesthesia care unit, which emphasizes the importance of its prevention.

The aim of this study is to investigate the effect of sugammadex vs. a conventional acetylcholinesterase inhibitor, neostigmine on emergence delirium (ED) during sevoflurane-rocuronium anesthesia in pediatric patients Additionally, the efficacy features of sugammadex compared to neostigmine will be examined by measuring the time from start of administration of reversal agents to recovery of TOF ratio to 0.7, 0.8, and 0.9.

Although the etiology of ED remains unclear, a sense of suffocation or breathing difficulty during emergence from anesthesia has been suggested as a possible cause. Thus, reversal of neuromuscular blockade with sugammadex in pediatric patients maintained with sevoflurane-rocuronium anesthesia may decrease ED due to its faster reversal of neuromuscular blockade and decreased possibility of residual blockade.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist (ASA) physical status I or II, preschool children scheduled for an elective tonsillectomy with or without adenoidectomy will be included in the study.

Exclusion Criteria:

* Patients will be excluded in cases of emergency surgery, developmental, psychological, cognitive or communication disorders, known or suspected neuromuscular disorders that may impair neuromuscular blockade, significant renal or hepatic dysfunction, coagulation disorders, family history of malignant hyperthermia, allergy to any of the drugs included in the study protocol, or usage of medication known to interact with rocuronium or sugammadex.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Kyun Kim, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Plaud B, Meretoja O, Hofmockel R, Raft J, Stoddart PA, van Kuijk JH, Hermens Y, Mirakhur RK. Reversal of rocuronium-induced neuromuscular blockade with sugammadex in pediatric and adult surgical patients. Anesthesiology. 2009 Feb;110(2):284-94. doi: 10.1097/ALN.0b013e318194caaa. PMID 19194156
- [Background] Locatelli BG, Ingelmo PM, Emre S, Meroni V, Minardi C, Frawley G, Benigni A, Di Marco S, Spotti A, Busi I, Sonzogni V. Emergence delirium in children: a comparison of sevoflurane and desflurane anesthesia using the Paediatric Anesthesia Emergence Delirium scale. Paediatr Anaesth. 2013 Apr;23(4):301-8. doi: 10.1111/pan.12038. Epub 2012 Oct 9. PMID 23043512
- [Background] Pieters BJ, Penn E, Nicklaus P, Bruegger D, Mehta B, Weatherly R. Emergence delirium and postoperative pain in children undergoing adenotonsillectomy: a comparison of propofol vs sevoflurane anesthesia. Paediatr Anaesth. 2010 Oct;20(10):944-50. doi: 10.1111/j.1460-9592.2010.03394.x. Epub 2010 Aug 24. PMID 20735801

RESULTS

PARTICIPANT FLOW:
Groups:
- Sugammadex: reversal of neuromuscular blockade with sugammadex
  Sugammadex Injection [Bridion]: Return to T2 point (two contractions) on TOF device is replied by iv 2 mg/kg sugammadex administration, contained in a blinded syringe.
- Neostigmine: reversal of neuromuscular blockade with neostigmine & glycopyrrolate
  Neostigmine+Glycopyrronium: Return to T2 point (two contractions) on TOF device is replied by iv 0.06 mg/kg neostigmine and 0.005 mg/kg glycopyrrolate administration, contained in a blinded syringe.
Period: Overall Study
Arm/Group | Sugammadex | Neostigmine
Started | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: One patient in Neostigmine group was dropped for the violation of protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex | Neostigmine | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.9 (1) | 5.5 (1.2) | 5.5 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 10 | 10 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 20 | 19 | 39
Region of Enrollment [Number; unit: participants]
  South Korea | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Pediatric Anesthesia Emergence Delirium Score
Description: Maximum Pediatric Anesthesia Emergence Delirium (PAED) score after arrival in the PACU.Higher values represent more emergence delirium (worse) PAED Score is represented with total PAED score summed up of subscales. The total score is reported and it ranges from 0 to 20. Higher score means worse state.
Time Frame: within 30 minutes after arrival at post-anesthesia care unit (PACU)
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 20 | 19
units on a scale | 18 [12.5 to 20] | 18 [9.5 to 20]

2. Secondary Outcome: Time Recovery of TOF Ratio to 0.7
Description: Time from the start of administration of reversal agents to recovery of the TOF ratio to 0.7
Time Frame: Time from the start of administration of reversal agents to recovery of the TOF ratio to 0.7, assessed up to 60 minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 20 | 19
seconds | 72.7 (37.7) | 167.4 (68.6)

3. Secondary Outcome: Time to Regular Breathing
Description: time from administration of reversal agent to time of deep, regular breathing
Time Frame: time from administration of reversal agent to time of deep, regular breathing, assessed up to 60 minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 20 | 19
seconds | 273.8 (147.4) | 345.1 (214.6)

4. Secondary Outcome: Time to Awakening
Description: time from administration of reversal agent to time of eye opening or child showing purposeful movement
Time Frame: time from administration of reversal agent to time of eye opening or child showing purposeful movements, assessed up to 60 minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 20 | 19
seconds | 275.8 (134.6) | 371.2 (195.1)

5. Secondary Outcome: Time to Extubation
Description: time from administration of reversal agent to time of tracheal extubation
Time Frame: time from administration of reversal agent to time of tracheal extubation, assessed up to 60 minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 20 | 19
seconds | 312.1 (155.0) | 427.3 (184.0)

6. Secondary Outcome: Time Recovery of TOF Ratio to 0.8
Description: Time from the start of administration of reversal agents to recovery of the TOF ratio to 0.8
Time Frame: Time from the start of administration of reversal agents to recovery of the TOF ratio to 0.8, assessed up to 60 minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 20 | 19
seconds | 83.9 (42.7) | 213.6 (81.8)

7. Secondary Outcome: Time Recovery of TOF Ratio to 0.9
Description: Time from the start of administration of reversal agents to recovery of the TOF ratio to 0.9
Time Frame: Time from the start of administration of reversal agents to recovery of the TOF ratio to 0.9, assessed up to 60 minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Sugammadex | Neostigmine
Number analyzed (Participants) | 20 | 19
seconds | 99.6 (38.2) | 253.1 (128.5)

ADVERSE EVENTS:
Time Frame: Anaphylaxis, bradycardia, vomiting, pain, nausea, hypotension, and headache are monitored at post-anesthetic care unit until the patients discharge. It took 1 hour after administration.
Arm/Group | Sugammadex | Neostigmine
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT03229486/Prot_SAP_001.pdf